CLINICAL TRIAL: NCT01878903
Title: Prospective Comparative Study of Electronic Visual Analogue Scale and Verbal Numerical Rating Scale in Acute Post-operative Pain.
Brief Title: Electronic Visual Analogue Scale in Acute Postoperative Pain
Status: Completed | Type: Observational
Sponsor: Cheung Chi Wai (Other)
Responsible Party: Sponsor-Investigator, Cheung Chi Wai, Clinical Associate Professor, The University of Hong Kong
Organization: The University of Hong Kong (Other)
Other Study IDs: UW-13-166
Record Dates: First submitted 2013-04-01; First posted 2013-06-17 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- i-pad VAS: All patients will be in one arm and they will be asked for post-operative pain using verbal NRS and visual VAS with i-pad
  Interventions: Other: Electronic VAS

INTERVENTIONS:
Other: Electronic VAS — Post-opearive pain patients will be assessed using electional VAS and verbal NRS
  Other Names: i-pad assessment

SUMMARY:
When assessing acute post-operative pain, the validity, reproducibility and reliability of Visual Analogue Scale (VAS) and verbal Numerical Rating Scale (NRS) have been investigated extensively. The use of electronic version of VAS has been published in the recent 10 years yet publication related to its use in pain medicine were few. Jamison et al have shown good correlation between electronic VAS vs paper VAS on healthy volunteers using weight as the stimulus. In normal subjects as well as fibromyalgia patients, electronic form of VAS could be used to describe different levels of experimental heat stimulation.

Long term study had been done where electronic pain diary were compared against paper diary in recording pain in 36 patients with chronic low back pain. The 2 scales showed good correlation. This author use a software that is Palm-top computer based. Following these few studies, validation study in chronic pain patient were published. A Palm-top computer based VAS was compared with paper NRS in 200 chronic pain patients. The pain level recorded by the two methods were considered equivalent by the author. However, Palm-top computer has almost disappeared from the market nowadays.

Recent handheld electronic devices (iPad®) were incorporated with touch screen input interface which allow users to use their finger as the input device. To our knowledge, there is no published data concerning iPad-based VAS, especially in post-operative pain. We would like to compare the data obtained from electronic VAS on iPad with verbal numerical rating scale when acute post-operative pain is assessed.

Hypothesis The null hypothesis is that the two pain measurement method do not correlate. The Spearman correlation coefficient between electronic VAS and verbal NRS will be reported.

DETAILED DESCRIPTION:
Objective:

To assess the agreement between the pain level measured by electronic VAS and verbal NRS in acute pain situation. Secondary objective is to determine the test-re-test reliability of electronic VAS.

Method:

All Chinese or English speaking patients 18 years or above, who are taken care by the acute pain service in Queen Mary Hospital are eligible for inclusion. Patients suffer from dementia, visual or hearing impairment will be excluded. Written consent will be obtained.

Pain specialist responsible for the acute pain service will assess patients' condition during daily ward round while patients are using patient controlled analgesia (PCA) device, receiving epidural infusion or peripheral nerve local anaesthetic infusion. For the pain assessment, patient will be asked to rate their current pain level using verbal numerical rating scale (NRS) as a standard or care. (0 being no pain, 10 being worst pain imaginable) Within one minute, the patient will be asked by the investigator, who is blinded to the verbal NRS, to rate the current pain level again on an electronic version of visual analogue scale on iPad® (vasQ Clinical©, Maki NAKATA 2011) The electronic VAS displayed on iPad® is a horizontal scale with "No Pain" on the left, "Worst Pain Imaginable" on the right. Patient can use the finger to mark the level of pain on the iPad® screen by moving a diamond shape marker alone the horizontal line. The length of the scale is divided electronically into 100 equal parts. There will be 101 possible score (0 - 10.0, which indicate the distance of the diamond marker from the left end of the scale. The score will be stored together with the patient's identifier.

Patients' clinical pain management will not be altered by the data obtained from the electronic VAS.

Patients will be asked to rate the current pain level after 1 minute using the electronic VAS again to evaluate the test-retest reliability of the tool.

Sample size Previous studies have shown that when VAS assessment was repeated in a short period of time, the standard deviation of the difference between the two measurements is around 8 mm (on a 100 mm scale). A sample size of 84 patients will be able to limit the 95% confidence interval of the mean difference between the pain assessment to +/- 3 mm. 92 patients will be recruited assuming a drop out rate of 10%.

Analysis The agreement between electronic VAS and verbal NRS will be evaluated using Spearman rank correlation6 and Bland-Altman method. The Spearman coefficient will be presented together with 95% confident interval (CI). The Bland-Altman method involves plotting the mean of the electronic VAS and NRS against the difference between the 2 scores for each pair of data. Mean difference +/- standard deviation of the differences between electronic VAS and verbal NRS will be presented.

The analysis will be repeated for the 2 sets of electronic VAS obtained 1 minute apart to evaluate the test-retest reliability of the electronic VAS.

ELIGIBILITY:
Inclusion Criteria:

* All Chinese or English speaking patients 18 years or above, who are taken care by the acute pain service in Queen Mary Hospital, Hong Kong are eligible for inclusion.

Exclusion Criteria:

* Patients suffer from dementia, visual or hearing impairment will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted at the population of Hong Kong.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2013-04; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Scores | The participants will be ask for pain scores (NRS and VRS with i-Pad) at postoperative day 1(the following day after the operation)

CONTACTS AND LOCATIONS:
Overall Officials: Chun Yin Wat, MBBS, Principal Investigator — Department of Anaesthesiology, Queen Mary Hospital, Hong Kong
Locations (1):
- Deaprtment of Anaesthesiology, The University of Hong Kong, Hong Kong, China